CLINICAL TRIAL: NCT05899491
Title: Role of ARMA in Selective Subset of Refractory GERD Patients- A Randomized Sham Control Trial.
Brief Title: Role of ARMA in Selective Subset of Refractory GERD Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARMA
Record Dates: First submitted 2023-04-01; First posted 2023-06-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2023-06

CONDITIONS: GERD; Reflux; Reflux Esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis, Peptic

STUDY DESIGN:
Intervention Model Description: A Randomized Sham Control Trial
Masking Description: A Randomized Sham Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARMA Group (Active Comparator): All patients in this group will undergo Anti-reflux mucosal ablation using upper gastrointestinal endoscopy. The stomach will be insufflated with CO2 to visualize the cardia in retroflex view.
  Interventions: Procedure: ARMA
- Sham Group (Sham Comparator): UGI Endoscopy will be performed under Propofol based sedation with scope kept inside for at least 5 minutes.
  Interventions: Procedure: UGI Endoscopy

INTERVENTIONS:
Procedure: ARMA — Patients will be instructed to fast for 6 hours pre-ARMA, the Procedure will be performed under propofol-based sedation. Patients will be in the left lateral decubitus position. The stomach will be insufflated with CO2 to visualize the cardia in retroflex view.
  Arms: ARMA Group
Procedure: UGI Endoscopy — UGI Endoscopy will be performed under propofol based sedation with scope kept inside for atleast 5 minutes.
  Follow up will include objective evaluation of reflux disease with: upper endoscopy, esophageal manometry, pHmetry, reflux questionnaire.
  Arms: Sham Group

SUMMARY:
To study the role of a novel endoscopic treatment technique (ARMA) in GERD patients who doesn't respond to PPI therapy (Proton Pump Inhibitor).

DETAILED DESCRIPTION:
Patients coming with symptoms of Gastroesophageal reflux disease (GERD) - A digestive disease in which stomach acid or bile irritates the food pipe lining, will be screened for eligibility and informed written consent will be taken. At initial screening, score based on clinical symptoms i.e. Gastroesophageal Reflux Disease- Quality of Life score (GERD HRQL) & Frequency Scale for the Symptoms of Gastroesophageal Reflux Disease Questionnaire (FSSG) score will be completed. All patients will undergo esophagogastroscopy (procedure to diagnose and treat problems in your upper GI (gastrointestinal) tract). to look for reflux (the backward flow of stomach acid into the tube that connects your throat to your stomach (esophagus)) related changes in the esophagus.

Esophageal high-resolution Manometry (procedure to diagnose and treat problems in your upper GI (gastrointestinal) tract) will be done to measure the various parameters which help doctor understand your disease.

24-hr pH impedance (procedure to diagnose and treat problems in your upper GI (gastrointestinal) tract) will be done after stopping anti-secretory medicines (medicines for the long-term treatment of GERD) for atleast three days to assess for esophageal parameters.

All patients will be divided randomly into two arms, ARMA and sham. Those in the ARMA arm will receive ARMA procedure, while patients in the sham arm will receive only upper gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Normal Upper Gastrointestinal endoscopy And
* 24 hour pH Impedance: AET < 6%, More than 80 refluxes
* Patients who are willing to give consent for the procedure

Exclusion Criteria:

* Large Hiatal hernia >3cm
* Lower esophageal sphincter (LES) pressure >15 mm Hg
* Paraesophageal hernia
* GE flap valve grade IV (Hill's classification)
* Barretts esophagus
* Esophageal dysmotility
* ASA physical status >II
* Previous esophageal or gastric surgery
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Improvement in Gastro esophageal reflux disease symptoms by more than 50% from baseline at 3 months. | One Year
  Improvement in Gastroesophageal reflux disease symptoms by more than 50% from baseline at 3 months which would be assessed based on visual analog scale VAS 0 LOW SCORE 10 WORSE SYMPTOM SCORE.

SECONDARY OUTCOMES:
Improvement in esophageal acid exposure | One Year
  Improvement in esophageal acid exposure in PH impedence monitoring report from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Singla, MD, Principal Investigator — Asian Institute of Gastroenterology, Hyderabad; Digvijay Chavan, Study Chair — Asian Institute of Gastroenterology, Hyderabad
Locations (1):
- Asian institute of Gastroenterology, hyderabad, India, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inoue H, Tanabe M, de Santiago ER, Abad MRA, Shimamura Y, Fujiyoshi Y, Ueno A, Sumi K, Tomida H, Iwaya Y, Ikeda H, Onimaru M. Anti-reflux mucosal ablation (ARMA) as a new treatment for gastroesophageal reflux refractory to proton pump inhibitors: a pilot study. Endosc Int Open. 2020 Feb;8(2):E133-E138. doi: 10.1055/a-1031-9436. Epub 2020 Jan 22. PMID 32010745
- [Background] Chou CK, Chen CC, Chen CC, Wu JF, Liao WC, Chiu HM, Wang HP, Wu MS, Tseng PH. Positive and negative impact of anti-reflux mucosal intervention on gastroesophageal reflux disease. Surg Endosc. 2023 Feb;37(2):1060-1069. doi: 10.1007/s00464-022-09605-z. Epub 2022 Sep 15. PMID 36109362
- [Background] Rodriguez de Santiago E, Albeniz E, Estremera-Arevalo F, Teruel Sanchez-Vegazo C, Lorenzo-Zuniga V. Endoscopic anti-reflux therapy for gastroesophageal reflux disease. World J Gastroenterol. 2021 Oct 21;27(39):6601-6614. doi: 10.3748/wjg.v27.i39.6601. PMID 34754155